CLINICAL TRIAL: NCT02878642
Title: Cohort Study to Assess Electronic-caps Defined Adherence Patterns - Virological Outcome Relationship Amongst HIV-1 Infected Subjects Receiving Dolutegravir-Based Antiretroviral Therapy)
Brief Title: Adherence to Dolutegravir and Outcome
Acronym: DOLUTECAPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 13-184
Record Dates: First submitted 2016-05-27; First posted 2016-08-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main assumption is that the dolutegravir can get virologic suppression to suboptimal adherence levels (between 80 and 95%, and after treatment interruptions) where other molecules are not capable, due to their pharmacokinetic/pharmacodynamic (pardonnance).

While the investigators goal is not to compare molecules (study with one arm) in terms of forgiveness, the results of this cohort in terms of forgiveness could be compared to other cohorts available.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1
* Age over 18 years
* Information letter signed
* ART (antiretroviral therapy) with at least 3 active molecules
* Patients starting treatment with dolutegravir (naïve to antiretroviral treatment, switch, virologic failure)

Exclusion Criteria:

* pregnant woman
* HIV-2
* Patient does not have responsibility for the observance of treatment (disorder of judgment, guardianship, institutionalization)
* Patient receiving aid incompatible with compliance with the use of electronic pillbox

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with HIV-1 treated with dolutegravir at week 16 and week 24
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12

PRIMARY OUTCOMES:
Adherence to dolutegravir measured by the electronic pill boxes | From baseline up to week 24
  Calculating the total compliance
Virologic Efficacy | week 24
  Are defined as secondary virological failure condition patients to S24 a viral load above 40 copies / ml on 2 consecutive samples.

SECONDARY OUTCOMES:
Patient Genotype resistance if failure | Week 16 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France